CLINICAL TRIAL: NCT05952544
Title: Does Protein Restriction Plus Essential Amino Acids and Keto-analogues Supplementation Have a Beneficial Effect on GFR Decline in CKD Patients?
Brief Title: Effect of Protein Restriction Plus EAA/KA Supplementation on GFR Decline in CKD
Status: Completed | Type: Observational
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Mohamed Mamdouh Mahmoud Mohamed Elsayed , MD, Lecturer, Alexandria University
Other Study IDs: effect of EAA/KA on GFR in CKD
Record Dates: First submitted 2023-07-01; First posted 2023-07-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Chronic Kidney Diseases
Keywords: protein restriction; essential amino acids; ketoanalogues; GFR; CKD
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Amino Acids, Essential; Diet, Protein-Restricted

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control group: include patients who were on low protein diet only
  Interventions: Other: low protein diet
- interventional group: include patients who consumed KA/EAA plus very low protein diet
  Interventions: Drug: essential amino acids and keto-analogues supplementation

INTERVENTIONS:
Drug: essential amino acids and keto-analogues supplementation — very low protein diet plus essential amino acids and keto-analogues supplementation
  Groups: interventional group
Other: low protein diet — patients were on low protein diet only
  Groups: control group

SUMMARY:
This study aims to investigate the effect of protein restriction plus KA/EAA supplementation on GFR decline in CKD patients.

DETAILED DESCRIPTION:
In chronic kidney disease (CKD) patients, ketoacid analogues of essential amino acids (KA/EAA) are administered to reduce the production of harmful metabolic products and enhance nutritional status. Protein restriction combined with AA supplement may have beneficial effects on CKD in several ways, by reducing nitrogen waste, oxidative stress, and inflammation, and by protecting against hemodynamic changes in glomerular hyperfiltration.

several clinical trials have documented that very low protein diets (VLPD) supplemented with KA/EAA preserve the rate of progression of advanced CKD. However, in long-term follow-up of the MDRD study, VLPD plus KA/EAA treatment did not delay progression to dialysis or transplantation.

As a result, no firm conclusions have been drawn on the effectiveness of protein-restricted diets combined with KA/EAA supplements in retarding CKD progression.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CKD stages (G2 to G4), aged ≥ 18 years old

Exclusion Criteria:

1. Active malignancy
2. Protein energy wasting
3. Advanced organ disease
4. pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: medical records of Patients with CKD stages (G2 to G4), will be retrospectively screened from December 2021 till December 2023.
  Patients will be divided into two groups:
  Control group who was on low protein diet only, while the other group (interventional) consumed KA/EAA plus very low protein diet.
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2023-07-20 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
GFR decline | 24 months
  effect on GFR change at one year from baseline in CKD patients

SECONDARY OUTCOMES:
effect on albumin | 24 months
  measurement of albumin change at one year from baseline
effect on calcium | 24 months
  measurement of calcium change at one year from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Mamdouh Elsayed, MD, Principal Investigator — lecturer; Bassant Sabry, Study Chair — pharmacist; Alaa Soliman, Study Chair — pharmacist; Mohamed A. Mekawy, Study Chair — pharmacist; Engy Emam, Study Chair — Clinical Pharmacist
Locations (1):
- Faculty of Medicine, Aexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Feiten SF, Draibe SA, Watanabe R, Duenhas MR, Baxmann AC, Nerbass FB, Cuppari L. Short-term effects of a very-low-protein diet supplemented with ketoacids in nondialyzed chronic kidney disease patients. Eur J Clin Nutr. 2005 Jan;59(1):129-36. doi: 10.1038/sj.ejcn.1602050. PMID 15354199
- [Background] Gao X, Huang L, Grosjean F, Esposito V, Wu J, Fu L, Hu H, Tan J, He C, Gray S, Jain MK, Zheng F, Mei C. Low-protein diet supplemented with ketoacids reduces the severity of renal disease in 5/6 nephrectomized rats: a role for KLF15. Kidney Int. 2011 May;79(9):987-96. doi: 10.1038/ki.2010.539. Epub 2011 Jan 19. PMID 21248717
- [Background] Jiang Z, Zhang X, Yang L, Li Z, Qin W. Effect of restricted protein diet supplemented with keto analogues in chronic kidney disease: a systematic review and meta-analysis. Int Urol Nephrol. 2016 Mar;48(3):409-18. doi: 10.1007/s11255-015-1170-2. Epub 2015 Nov 30. PMID 26620578
- [Background] Menon V, Kopple JD, Wang X, Beck GJ, Collins AJ, Kusek JW, Greene T, Levey AS, Sarnak MJ. Effect of a very low-protein diet on outcomes: long-term follow-up of the Modification of Diet in Renal Disease (MDRD) Study. Am J Kidney Dis. 2009 Feb;53(2):208-17. doi: 10.1053/j.ajkd.2008.08.009. Epub 2008 Oct 31. PMID 18950911